CLINICAL TRIAL: NCT07091903
Title: The Effect of Diaphragmatic Breathing Exercises Applied in Addition to Conventional Treatment on Pain, Upper Extremity Stability, and Anxiety in Individuals With Rotator Cuff Lesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Zeynep HOŞBAY, Professor, Physiotherapist, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Breath in rotator cuff lesion
Record Dates: First submitted 2025-07-15; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Rotator Cuff Lesions
Keywords: Rotator Cuff Lesions; Anxiety; Diaphragmatic Breathing Exercise; Pain; Upper Extremity Stability
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical Trial
Who Masked: Participant
Masking Description: Participants does not know which type of treatment is received themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Respiratory Group (Experimental): Diaphragmatic breathing exercises in addition to conventional physiotherapy and post-isometric relaxation technique were applied to the respiratory group.
  Interventions: Other: Diaphragmatic breathing exercise; Other: Conventional physiotherapy and post-isometric relaxation technique
- The Control Group (Experimental): Conventional treatment and post-isometric relaxation technique were applied to the control group.
  Interventions: Other: Conventional physiotherapy and post-isometric relaxation technique

INTERVENTIONS:
Other: Diaphragmatic breathing exercise — Individuals in the respiratory group received a physiotherapy and rehabilitation program for 6 weeks, 3 days a week. Diaphragmatic breathing exercise was performed with the participants in a supine position with bent knees, 10 repetitions and 3 sets.
  Arms: The Respiratory Group
Other: Conventional physiotherapy and post-isometric relaxation technique — Individuals in the respiratory group received a physiotherapy and rehabilitation program for 6 weeks, 3 days a week. The treatment of individuals in this group included conventional physiotherapy and post-isometric relaxation technique. Conventional treatment included an exercise program consisting of Wand, Codman, and finger ladder exercise, in addition to 20 min HotPack, 20 min TENS and 5 min Ultrasound modalities. Each of the exercises was applied as 10 repetitions and 1 sets. Post-isometric relaxation technique was applied with 5 seconds of isometric contraction in the direction of flexion, abduction, internal and external rotation, 5 repetitions, 2 sets.

SUMMARY:
The goal of this study is to investigate the effects of diaphragmatic breathing exercises in addition to conventional treatment and post isometric relaxation technique on pain, range of motion, functionality, upper extremity stability, and anxiety in individuals with rotator cuff lesions. The study included 32 participants aged between 18 and 65 years, diagnosed with rotator cuff lesions. The control group (n=16) received conventional treatment and the post-isometric relaxation technique, while the respiratory group (n=16) received diaphragmatic breathing exercises in addition to conventional treatment and the post-isometric relaxation technique. The researcher used the Visual Analog Scale (VAS) to assess pain intensity, a universal goniometer to measure range of motion, the Shoulder Pain and Disability Index (SPADI) to evaluate functional status, the Upper Extremity Y-Balance Test to assess upper extremity stability, the State-Trait Anxiety Inventory (STAI) to measure anxiety levels, and a finger-type pulse oximeter to record pulse and oxygen saturation values. The researcher used SPSS V.27 program for statistical analysis of the data.

DETAILED DESCRIPTION:
Shoulder pain is a common musculoskeletal problem affecting a large portion of the general population. Its prevalence ranges from 7% to 25%. One of the most common causes is rotator cuff lesions. Rotator cuff lesions are pathologies that begin with acute tendonitis and progress to partial or full-thickness ruptures as degeneration progresses, leading to extensive progression. Their prevalence among individuals with shoulder pain exceeds 70%. Studies have shown that the incidence increases after age 40, and this rate exceeds 50% in those over age 60. The most common clinical symptoms observed in patients with rotator cuff lesions are decreased shoulder range of motion and flexibility, pain, and impaired shoulder function. This resulting pain and loss of function significantly impact performance in activities of daily living and quality of life. The literature indicates that patients with rotator cuff lesions generally experience additional problems such as depression, anxiety, poor sleep quality, and kinesiophobia. Psychological factors are also thought to play a role in the etiology and chronicity of shoulder pain. In order to achieve a functional movement, parameters such as sufficient November muscle strength, mobility, stability, flexibility, coordination, balance are required along the basic movement pattern. In shoulder pathologies, decreased mobility due to restriction of upper limb movement affects stability. The deterioration of these components leads to a deterioration of functional movement. Conservative or surgical methods can be used in the treatment of rotator cuff lesions. Conservative treatment is known to be the preferred and effective method. Nonsteroidal anti-inflammatory drugs, corticosteroid injections, activity modification, and physiotherapy constitute conservative treatment. Physiotherapy includes rest, stretching, manual therapy, active and passive shoulder exercises, and physical therapy modalities. The primary goals of the treatment program are to reduce pain and dysfunction, regain range of motion by stretching the posterior capsule and other soft tissues, and increase rotator cuff and scapular muscle strength. Post-isometric relaxation is a muscle energy technique (MET) defined as the reduction of tone in the agonist muscle after isometric contraction. It is considered a manual therapy technique, aims to reduce muscle tension by regulating muscle function, and is used in both subacute and chronic settings. Muscle energy techniques have been found to have a positive effect in reducing pain and increasing range of motion in patients with adhesive capsulitis and impingement. Diaphragmatic breathing exercises contribute to core stabilization. Diaphragmatic movements during respiration affect the sympathetic and parasympathetic nervous systems. Recent studies have shown that breathing exercises are among the pain-reducing interventions. Pro-inflammatory markers are reduced with breathing exercises, thus demonstrating their effectiveness in reducing inflammation. Relaxation and deep breathing exercises are believed to reduce pain and improve quality of life in individuals with shoulder pain. Furthermore, breathing exercises and breath awareness enhance psychological and physical well-being and, through the resulting relaxation effect, reduce pain. There are studies demonstrating that diaphragmatic breathing exercises positively impact trunk muscle activity and functional levels in musculoskeletal conditions such as low back pain. Proprioceptive neuromuscular facilitation and breathing exercises applied to patients with frozen shoulder have been shown to reduce pain and increase range of motion. Similarly, diaphragmatic mobilization and diaphragmatic breathing exercises have been found to be effective in reducing pain and improving quality of life in individuals with shoulder pain. A review of the literature reveals a limited number of studies investigating the effectiveness of diaphragmatic breathing exercises in shoulder patients. No studies have been found evaluating the effects of diaphragmatic breathing exercises applied in addition to post-isometric relaxation techniques on upper extremity stability and anxiety parameters in individuals with rotator cuff lesions. The aim of our study was to investigate the effects of diaphragmatic breathing exercises applied in addition to conventional treatment and post-isometric relaxation techniques on pain, range of motion, functionality, upper extremity stability, and anxiety parameters in individuals with rotator cuff lesions.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18 and 65 years of age,
* Having been diagnosed with a rotator cuff lesion,
* Having unilateral shoulder pain that has persisted for at least 4 weeks,
* Having no cognitive or mental problems,
* Individuals who are willing to participate in the study and are willing to cooperate.

Exclusion Criteria:

* Patients who have received local corticosteroid injections or corticosteroid treatment within the last three months,
* Patients who have a total rotator cuff tear (Stage 3 according to Neer),
* Patients who have shoulder instability or fractures,
* Patients who have a history of shoulder, upper extremity, or thoracic surgery,
* Patients who have neuromuscular disease, unstable angina, malignancy, pulmonary or vascular problems, inflammatory arthritis, vertigo, various vestibular system pathologies, and communication problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-06-10 (Actual)

PRIMARY OUTCOMES:
Range of Motion of the Shoulder Joint | 6 weeks
  In our study, individuals' shoulder joint range of motion was measured with a "universal goniometer" and evaluated. Goniometric measurement is an objective method frequently used in ROM evaluation. Before and after treatment, individuals' shoulder flexion, extension, abduction, external rotation and internal rotation active range of motion was measured with a universal goniometer. Measurements were made 3 times and the average of each measurement was recorded.
Shoulder Pain | 6 weeks
  In our study, pain was assessed using the Visual Analog Scale (VAS). The Visual Analog Scale is a scale in which pain intensity is expressed by marking on a line 0-10 cm long. Before the assessment, participants were informed that the numbers on the scale were expressed as "'0: no pain' and '10: unbearable pain'" and were asked to mark the intensity of pain they felt at rest, during activity, and at night on the line.
Shoulder Functionality | 6 weeks
  Patients' functionality was assessed with the Shoulder Pain and Disability Index (SPADI). The index was developed to measure pain and disability. It contains 5 questions for pain and 8 questions for disability. Patients are asked to answer each question on a scale from 0 to 10 (0 = no pain/strain; 10 = maximum pain experienced/inability to do anything). The score is calculated separately for pain, disability, and total score. The score is calculated by adding the scores for each section, dividing by the maximum possible score for that section, and multiplying by 100. Higher scores indicate greater pain and disability.
Anxiety | 6 weeks
  The State-Trait Anxiety Inventory (STAI) was used to assess patients' anxiety levels. The original version of the scale was developed by Spielberger and colleagues. This self-assessment scale consists of two subscales: State and Trait Anxiety. State anxiety assesses an individual's level of anxiety in a given situation, while trait anxiety indicates an individual's tendency to experience anxiety. The scale consists of 40 items (20 for state anxiety and 20 for trait anxiety), and each item is scored from 1 to 4. The total score ranges from 20 to 80. Higher scores indicate higher anxiety levels.
Upper Extremity Stability and Mobility | 6 weeks
  The Y-Balance Test was used to assess patients' upper extremity stability and mobility. The upper extremity Y-Balance test is a functional test that allows simultaneous assessment of upper extremity stability, core stability, and contralateral upper extremity mobility. In the test, the subject stabilizes body weight with one upper extremity while maximally extending the other extremity in three directions. Due to the cost of the original Y-Balance Test kit, a modified Y-Balance test was used in our study. The farthest distance reached in each direction was recorded in cm. Three measurements were taken on the right and left arms. To eliminate the upper extremity length advantage, composite values were calculated for both the right and left extremities.
Pulse | 6 weeks
  Pulse oximetry is a non-invasive, painless, and reliable method for measuring oxygen saturation in arterial blood. Patients' pulse values were assessed using a finger-type pulse oximetry device.
Oxygen Saturation | 6 weeks
  Pulse oximetry is a non-invasive, painless, and reliable method for measuring oxygen saturation in arterial blood. Patients' oxygen saturation values were assessed using a finger-type pulse oximetry device.

CONTACTS AND LOCATIONS:
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee BK. Effects of the combined PNF and deep breathing exercises on the ROM and the VAS score of a frozen shoulder patient: Single case study. J Exerc Rehabil. 2015 Oct 30;11(5):276-81. doi: 10.12965/jer.150229. eCollection 2015 Oct. PMID 26535219
- [Background] Fernandez-Lopez I, Pena-Otero D, Atin-Arratibel MLA, Eguillor-Mutiloa M, Bravo-Llatas C, Genoves-Crespo M, Callejas-Gonzalez FJ. Effects of diaphragm muscle treatment in shoulder pain and mobility in subjects with rotator cuff injuries: A dataset derived from a pilot clinical trial. Data Brief. 2021 Feb 12;35:106867. doi: 10.1016/j.dib.2021.106867. eCollection 2021 Apr. PMID 33665260